CLINICAL TRIAL: NCT04242004
Title: Effects of Docosahexanoic Acid on Neurocognitive Impairment in HIV-infected Patients: A Randomized, Double-blind, Placebo-controlled Study
Brief Title: Effects of Docosahexanoic Acid on Neurocognitive Impairment in HIV-infected Patients
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB#2019-06-0759
Record Dates: First submitted 2020-01-14; First posted 2020-01-27 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Neurocognitive Impairment
Keywords: HIV-infected patients; neurocognitive impairment; gut microbiota; fatty acid docosahexaenoic; randomized controlled trial
MeSH Terms: interventions — Docosahexaenoic Acids; Capsules; Soybean Oil

STUDY DESIGN:
Intervention Model Description: Randomization (1:1) was performed according to a computer-generated random sequence, which was used to allocate the participants either to the dietary supplement or the placebo group.
Who Masked: Participant, Investigator
Masking Description: Participants, and investigators assessing outcome measures were blind to the intervention condition. Blinding was maintained until data analysis was completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DHA group (Experimental)
  Interventions: Drug: Docosahexaenoic acid (DHA) capsules
- placebo group (Placebo Comparator)
  Interventions: Dietary Supplement: Soy oil capsules

INTERVENTIONS:
Drug: Docosahexaenoic acid (DHA) capsules — Treatment was provided as 7 omega-3 fatty acid (Lovaza) capsules daily. Each capsule contained 1 g of omega-3 fatty acids with approximately 450 mg of docosahexaenoic acid (DHA).
  Arms: DHA group
Dietary Supplement: Soy oil capsules — The placebo was identical looking capsules that contained soy oil
  Arms: placebo group

SUMMARY:
Neurocognitive impairment (NCI) is one of the serious complications of elderly HIV-infected patients. The destruction of intestinal mucosal barrier and imbalance of bacterial flora caused by aging and HIV infection may be an important factor promoting the occurrence of NCI. Therefore, it is important to understand changes in gut microbiota of HIV-infected patients with NCI. Higher dietary intake of the essential fatty acid docosahexaenoic (DHA) has been associated with better cognitive performance in several epidemiological studies. To date, data are limited showing that DHA administration leads to benefits for behavioral disorders by modulating gut microbiota composition; the few studies on this subject, mostly completed in animal models. Moreover，low levels of DHA have been found in HIV-infected patients. The effect of DHA supplementation on gut microbiota and NCI status of HIV-positive patients have not been evaluated yet. Investigators aim to implement a case-control study to identify the relationship between gut microbiota and NCI in HIV-infected patients. At the meantime, investigators aim to implement a randomized, double-blind, placebo-controlled clinical trial to assess DHA supplementation in HIV-infected patients with NCI for 16 weeks. The effect of DHA on gut microbiota and NCI were evaluated. Also, investigators aim to identify if the benefits for NCI of DHA caused by modulating gut microbiota composition and metabolites.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients
* Age ≥18 years
* Established diagnosis of HIV-1 infection, under stable cART for the prior 6 months and throughout the study period
* Presence of neurocognitive impairment was assessed using the global deficit score (GDS), calculated as the average of deficit scores across all neuropsychological test. The cut-off for NCI was a GDS score ≥ 0.5

Exclusion Criteria:

* Age <18 years,
* BMI >30 kg/m2
* Pregnancy or lactation
* A history of diabetes mellitus, cardiovascular and cerebrovascular diseases, or serious diseases such as liver, kidney and hematopoietic system disease
* Known intolerance to n-3 PUFA preparations.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2019-10-30 (Actual); Primary Completion 2020-03-01 (Estimated); Study Completion 2020-05-01 (Estimated)

PRIMARY OUTCOMES:
Neurocognitive impairment | 16 weeks
  Participants underwent neurocognitive testing using an internationally validated comprehensive neurocognitive test battery covering 7 cognitive domains: verbal fluency, speed of information processing, executive functioning, learning, memory, attention/working memory and motor skills. Demographically-corrected (age, education, gender) T scores (mean of 50, standard deviation of 10) were developed based upon an age-matched control group. Individual test deficit scores, determined via demographically-adjusted T scores, ranged from 0 (T score of > 40) to 5 (T score < 20). Neurocognitive impairment (NCI) was assessed using the global deficit score (GDS), calculated as the average of deficit scores across all neuropsychological test. The cut-off for NCI was a GDS score ≥ 0.5
Gut microbiota | 16 weeks
  Investigators characterized the 16S rDNA fecal microbiome in participants. Shannon diversity index (SDI) was used to evaluate alpha (within sample) diversity. Beta (between sample) diversity was examined using principle coordinate analysis (PCoA) of unweighted Unifrac distances. Relative abundance of microbial taxa was compared between samples using Linear Discriminant Analysis Effect Size (LEfSe)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of epidemiology, School of public health, Fudan University,, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dong R, Lin H, Ding Y, Chen X, Shi R, Yuan S, Li J, Zhu B, Xu X, Shen W, Wang K, Ding D, He N. Effects of Docosahexanoic Acid on Gut Microbiota and Fecal Metabolites in HIV-Infected Patients With Neurocognitive Impairment: A 6-Month Randomized, Double-Blind, Placebo-Controlled Trial. Front Nutr. 2022 Jan 21;8:756720. doi: 10.3389/fnut.2021.756720. eCollection 2021. PMID 35127778